CLINICAL TRIAL: NCT04290598
Title: Clinical Effects of Dehydration on Tooth Colour: How Much and How Long?
Brief Title: Clinical Effects of Dehydration on Tooth Colour
Status: Completed | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Huseyin Hatirli, Assistant Professor, Tokat Gaziosmanpasa University
Other Study IDs: GaziosmanpasaU2019-46
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Color; Change Teeth, Posteruptive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Dental restorations should mimic sound tooth structures in terms of color and optical properties especially in the anterior region. However, closely matching natural teeth with a restoration can be one of the most challenging procedure in restorative dentistry. Shade matching includes color determination, color communication with dental lab and color reproduction with dental restoration for indirect techniques or color determination and selection of the appropriate material and application method when using direct techniques. Therefore color selection is the first critical step in the restoration procedures and should be carried out properly.

Color determination must be carried out before any of the restorative procedures, isolation or impression. Most of the dental procedures cause dehydration and increase the opacity of the enamel and teeth appear whiter. Few clinical and in vitro studies evaluated the degree of color change after dehydration and rehydration periods. However, inconsistencies exist between studies in terms of color change degree and duration of return to appreciable values.

The aim of the present study was to evaluate the degree of color change in half an hour dehydration period of the teeth and to determine if color return to baseline after half an hour or 24 hours.

According to the null hypotheses of the study:

* There is no perceptible difference occur after tooth dehydration.
* Tooth color will not return to baseline values after half an hour or 24 hours rehydration periods.

DETAILED DESCRIPTION:
Color measurements Color measurements were performed with a spectrophotometer (SpectroShade Micro, MHT Optic Research AG, Niederhasli, Switzerland) by the same experienced dentist in the present study. Spectrophotometer was calibrated and used according to manufacturer instructions before each set of measurements. All participants were asked for not to mouth breath during color measurements. All of the color measurements were carried out under standard light conditions with the aim of minimizing the possible inaccurate readings.

Dehydration procedure Spectrophotometric color measurements were performed at the study inception and baseline color parameters were recorded. Lips were retracted by using a lip and cheek retractor which placed within 10 s. Upper central and lateral incisors were isolated with cotton rolls and air dried for 5 s. Excess saliva was removed with a suction and participants keep their mouth half-opened with the help of silicone mouth bite blocks. Spectrophotometric measurements were carried out three times during 30 min with 10 min intervals during the dehydration period for each test tooth.

Rehydration procedure At the end of the dehydration procedure, lip retractor and cotton rolls were removed and full-mouth rinse with water was done for 30 s. Participants asked to drink a bottle of water and close their mouth for 30 min. Participants were asked to return to routine daily activity, but not to consume staining beverages such as coffe or red wine. Tooth rehydration process was started when test teeth get in contact with saliva. Spectrophotometric measurements were carried out at 30 min and 24 h of rehydration.

CIELAB color parameters (L*,a*,b*) were used to calculate color differences (ΔE) between baseline and other measurement periods for each tooth and gingival, middle and incisal thirds separetely. Color difference was calculated by using an equation; ΔE*=[(ΔL*)2+(Δa*)2+(Δb*)2]1/2. ΔE values were compared to threshold values of acceptability(ΔE*=3,7) and perceptibility(ΔE*=1). 11 Color difference and color parameters of 30 min and 24h dehydration was compared to baseline color parameters.

ELIGIBILITY:
Inclusion Criteria:

* To be in the age range of 18-45 years
* Upper central and lateral incisors should have a good periodontal condition and should be sound with no wear, restorations, internal or external discoloration

Exclusion Criteria:

* Recent fixed orthodontic appliance
* Vital tooth bleaching in the last year
* Medication, affecting salivary flow or complaint of dry mouth

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Participants will be selected amoung patients referring for dental treatments to Tokat Gaziosmanpasa University Faculty of Dentistry. Patients in the age range of 18-45 years and meeting inclusion criteria will be participated in this study.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-12-27 (Actual)

PRIMARY OUTCOMES:
Degree of color change after dehydration period | Thirty minutes dehydration period and rehydration period after 24 hours.
  CIELAB color system and L*,a*,b* parameters and delta E values

CONTACTS AND LOCATIONS:
Overall Officials: Huseyin Hatirli, Principal Investigator — assistant professor
Locations (1):
- Tokat Gaziosmanpasa University Faculty of Dentistry, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suliman S, Sulaiman TA, Olafsson VG, Delgado AJ, Donovan TE, Heymann HO. Effect of time on tooth dehydration and rehydration. J Esthet Restor Dent. 2019 Mar;31(2):118-123. doi: 10.1111/jerd.12461. Epub 2019 Feb 23. PMID 30801926
- [Background] Burki Z, Watkins S, Wilson R, Fenlon M. A randomised controlled trial to investigate the effects of dehydration on tooth colour. J Dent. 2013 Mar;41(3):250-7. doi: 10.1016/j.jdent.2012.11.009. Epub 2012 Nov 14. PMID 23160038
- [Background] Russell MD, Gulfraz M, Moss BW. In vivo measurement of colour changes in natural teeth. J Oral Rehabil. 2000 Sep;27(9):786-92. doi: 10.1046/j.1365-2842.2000.00610.x. PMID 11012854